CLINICAL TRIAL: NCT02636140
Title: Effect of Light Spectrum on Pupil Function
Brief Title: Color and Pupil Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jamie M. Zeitzer, Ph.D., Assistant Professor, VA Palo Alto Health Care System
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: IRB-36326
Record Dates: First submitted 2015-12-17; First posted 2015-12-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Pupil
MeSH Terms: interventions — Light

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Light (Experimental): Randomized amount and color of light
  Interventions: Other: Light

INTERVENTIONS:
Other: Light — A brief, 1 minute exposure to light of varying color and intensity. The combination of color and intensity will be the same in all participants, but the order in which they are received is randomized.

SUMMARY:
This study will examine the effects of different colors of light on pupil function and alertness.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-35
* Good health

Exclusion Criteria:

* Sleep disorder
* Extreme chronotype
* Smoker
* Abnormal color vision
* Ocular pathology (other than mild or moderate refractive error)
* Visual field defects
* Alcohol abuse
* Use of illegal drugs

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-02; Primary Completion 2016-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Change in pupil size | Baseline and 10 minutes
  Change in pupil size from baseline during and following brief light exposure